CLINICAL TRIAL: NCT00659061
Title: Monitoring and Evaluation of Micronutrients (Sprinkles) Project
Acronym: Sprinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Micronutrient Initiative (Other); M/S SEBCON (Other); Pakistan Ministry of Health (Other Government); National Programme of Family Planning and Primary Health Care (Unknown)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Founding Director, Centre of Excellence in Women and Child Health, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 754-Ped/ERC-07
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: micronutrients
MeSH Terms: conditions — Anemia | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Multiple micronutrient fortificant (Sprinkles) and nutrition education given by LHWs.
  Interventions: Dietary Supplement: SPRINKLES; Behavioral: Nutrition education
- Control (No Intervention): Routine public health massages by Lady Health Workers (LHWs) during their community visits.

INTERVENTIONS:
Dietary Supplement: SPRINKLES — Sprinkles is a multiple micronutrient fortificant. It is packed as a single serving sachets each containing micro encapsulated iron (12.5 mg), zinc (7.5 mg), vitamin C (30 mg), vitamin A (300 µg), vitamin D (5 µg), folic acid (150 µg) and iodine (90µg).
  Two month supply of the Sprinkle sachet along with advice on its benefits as well as its appropriate use will be given by the LHWs. The LHWs will also provide their age-appropriate nutritional advice as per their regular door to door community services.
  Other Names: Multiple micronutrient fortificant
  Arms: Intervention
Behavioral: Nutrition education — Nutrition education will be provided by LHWs as per their regular routine monthly door to door community services
  Arms: Intervention

SUMMARY:
The purpose of this study is 1) to evaluate the effectiveness in reducing anemia among children 6-24 months of age by providing daily micronutrient Sprinkles through the Government of Pakistan's Lady Health Worker program; 2) to assist in the monitoring the National Sprinkles Pilot Project.

DETAILED DESCRIPTION:
According to the recent National Nutrition Survey in Pakistan (2001-2002), approximately 66.5% of children under five have anaemia.

Looking at the magnitude of the problem, National Program for Family Planning (FP) and Primary Health Care (PHC) (also known as the Lady Health Workers (LHW) Program) has developed National Sprinkles Pilot Project Proposal with technical assistance of Micronutrient Initiative and Aga Khan University (AKU). As the projects technical partner, AKU is responsible to conduct the monitoring and evaluation of the project.

The study will use a cluster randomized pre-post intervention design that compares before and after hemoglobin (Hb) measurements, serum ferritin, serum retinol and urinary iodine among children who received Sprinkles and age-appropriate feeding advice (Sprinkles-Advice group) and children who only receive age-appropriate feeding advice (Advice-only group). Age-appropriate feeding advice is part of the standard nutrition messages given by all Lady Health Workers (LHWs) during their community visits. However, intervention LHWs, will give additional advice regarding the benefits of Sprinkles and its appropriate use.

The target population selected for the study consisted of children between the ages of six and eighteen months of age in the catchment area of the Lady Health Workers.

ELIGIBILITY:
Inclusion Criteria:

* Child's mother gives written consent after hearing an explanation of the study
* Random selection of child in household with more than one eligible child

Exclusion Criteria:

* Any household in which consent is not given
* Children with any congenital or physical disability (such as cleft palate, Down's Syndrome, etc.)
* Child from a family which intends to migrate during the study period

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 610 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, MD, PhD, Study Chair — Aga Khan University
Locations (1):
- AKU-Peds Naushero Feroze Site Office, Naushero Feroze, Sindh, Pakistan

RESULTS

PARTICIPANT FLOW:
Groups:
- Sprinkle-Advice: Sprinkles and age-appropriate feeding advice given by Lady Health Workers (LHWs). Age-appropriate feeding advice is part of the standard nutrition messages given by all Lady Health Workers (LHWs) during their community visits.
- Advice Only: Age-appropriate feeding advice given by LHWs as part of the standard nutrition messages given by all Lady Health Workers (LHWs) during their community visits.
Period: Overall Study
Arm/Group | Sprinkle-Advice | Advice Only
Started | 308 | 302
Completed | 287 (Those with either complete or partial biochemical and anthropometric data) | 287 (Those with either complete or partial biochemical and anthropometric data)
Not Completed | 21 | 15
Not completed — Migration due to political unrest | 21 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sprinkle-Advice | Advice Only | Total
Number analyzed (Participants) | 308 | 302 | 610
Age, Continuous [Mean (Standard Deviation); unit: months] | 12 (3.2) | 12.3 (3.3) | 12.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 155 | 327
  Male | 136 | 147 | 283

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anemia
Description: number with mild to severe anemia (hemoglobin(Hb)<11g/dL)
Time Frame: Baseline hemoglobin (Hb) taken at time of enrollment; Endline Hb taken 4-5 months post enrollment
Measure: Number; unit: participants
Arm/Group | Sprinkle-Advice | Advice Only
Number analyzed (Participants) | 287 | 284
participants
  Baseline anemia prevalence | 185 | 172
  Endline anemia prevalence | 139 | 191
Statistical Analysis 1: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.32, Chi-squared — at baseline
Statistical Analysis 2: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p < 0.001, Chi-squared — at endline

2. Secondary Outcome: Vitamin A Status of Participants - Post Intervention
Description: Categorized as <20ug/dL; 20-40 ug/dL; >40 ug/dl
Time Frame: Measurement taken 4-5 months post enrollment
Population: those who had endline assessment of serum vitamin A
Measure: Number; unit: participants
Arm/Group | Sprinkle-Advice | Advice Only
Number analyzed (Participants) | 232 | 232
participants
  Low (<20 ug/dl) | 74 | 115
  Moderate (20-40 ug/dl) | 96 | 89
  High (>40 ug/dl) | 62 | 28

3. Secondary Outcome: Mean Vitamin A Serum Retinol (ug]dl) Taken Post Intervention
Time Frame: Measurement taken 4-5 months post enrollment
Measure: Mean (95% Confidence Interval); unit: ug/dl
Arm/Group | Sprinkle-Advice | Advice Only
Number analyzed (Participants) | 277 | 275
ug/dl | 31.8 [28.4 to 35.2] | 25.1 [22.5 to 27.8]
Statistical Analysis 1: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p < 0.000, ANOVA; adjusted for baseline, child age, sex, number of sprinkles sachets consumed, number of mths between enrollment and endline Hb measurement)

4. Primary Outcome: Number of Participants With Moderate to Severe Anemia
Description: number of participants with moderate - severe anemia defined as Hb < 10g/dL
Time Frame: Baseline Hb taken at time of enrollment; Endline Hb taken 4-5 months post enrollment
Measure: Number; unit: participants
Arm/Group | Sprinkle-Advice | Advice Only
Number analyzed (Participants) | 287 | 284
participants
  Baseline | 114 | 102
  Endline | 84 | 138
Statistical Analysis 1: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.34, Chi-squared — baseline
Statistical Analysis 2: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p < 0.001, Chi-squared — endline

5. Primary Outcome: Mean Hemoglobin of Participants Post Intervention
Time Frame: Endline Hb taken 4-5 months post enrollment
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Sprinkle-Advice | Advice Only
Number analyzed (Participants) | 227 | 264
g/dL | 10.97 [10.7 to 11.3] | 9.98 [9.7 to 10.2]
Statistical Analysis 1: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.000, ANOVA — endline; adjusted for baseline child age, sex, # of sprinkle sachet consumed, # of mths between enrollment and endline Hb measurement

6. Secondary Outcome: Percentage of Underweight Participants
Description: Underweight defined as Weight for Age Z score < -2 standard deviation (SD)
Time Frame: Baseline measurements taken at time of enrollment; Endline measurements taken 4-5 months post enrollment
Population: those who had complete baseline anthropometric measures
Measure: Number; unit: percentage of participants
Arm/Group | Sprinkle-Advice | Advice Only
Number analyzed (Participants) | 285 | 286
percentage of participants
  Baseline Underwt % | 49 | 48
  Endline Underwt % | 35 | 44
Statistical Analysis 1: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.7, Chi-squared — baseline
Statistical Analysis 2: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.02, Chi-squared — endline

7. Secondary Outcome: Percentage of Participants With Stunted Growth
Description: Stunted defined as Height for Age Z-score < -2 standard deviation
Time Frame: Baseline measurements taken at time of enrollment; Endline measurments taken 4-5 months post enrollment
Population: Those who had complete anthropometric measurements at endline
Measure: Number; unit: percentage of participants
Arm/Group | Sprinkle-Advice | Advice Only
Number analyzed (Participants) | 286 | 287
percentage of participants
  Baseline Stunted % | 55 | 57
  Endline Stunted % | 62 | 61
Statistical Analysis 1: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.62, Chi-squared — baseline
Statistical Analysis 2: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.89, Chi-squared — endline

8. Secondary Outcome: Percentage of Participants With Wasted Growth
Description: Wasted defined as Weight for Height Z-score < -2SD
Time Frame: Baseline measurements taken at time of enrollment; Endline measurements taken 4-5 months post enrollment
Population: those who had complete anthropometric measurements at endline
Measure: Number; unit: percentage of participants
Arm/Group | Sprinkle-Advice | Advice Only
Number analyzed (Participants) | 284 | 286
percentage of participants
  Baseline Wasted % | 24 | 24
  Endline Wasted % | 13 | 15
Statistical Analysis 1: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.93, Chi-squared — baseline
Statistical Analysis 2: Comparison: Sprinkle-Advice vs Advice Only; Test type: Superiority or Other; p = 0.49, Chi-squared — endline

LIMITATIONS AND CAVEATS:
The attrition rate was high (6.8% in intervention group and 5.0% in the control group) due to unforeseen migration because of political unrest in the region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No